CLINICAL TRIAL: NCT07109635
Title: A Post Market Non-Interventional Study of Safety and Performance of RefillHA Volume+, a Dermal Filler for Facial Soft Tissue Augmentation and Correction of Facial Wrinkles and Folds
Brief Title: Post Market Study of Safety and Performance of RefillHA Volume+ for Facial Soft Tissue Augmentation and Correction of Wrinkles and Folds
Status: Completed | Type: Observational
Sponsor: Glyance (Industry)
Responsible Party: Sponsor
Other Study IDs: PMCF-SP-200-02
Record Dates: First submitted 2025-07-24; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Wrinkles Such as Nasolabial Folds
Keywords: wrinkles

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects over the age of 18 who are seeking correction of facial wrinkles and folds and/or soft tiss

SUMMARY:
This post market study was designed to collect clinical data regarding the safety and performance of RefillHA Volume+ upon its launch, from patients treated with the product in a routine clinical setting of treatments.

In this study, patients seeking correction of facial wrinkles and folds and/or soft tissue augmentation who are candidates for treatment with RefillHA Volume+ according to its approved use will be offered to participate in the study. Eligible patients who are willing to participate in the study, after signing an informed consent, will be treated with RefillHA Volume+ in the facial regions where correction is requested, subject to the advice of the treating physician and in accordance with the approved use.

After recieving initial treatment, participants will attend 2 to 4 in-clinic follow-up visits, during which they will be eligible to receive additional treatment with RefillHA Volume+ (up to two additional treatments during the follow-up period) if, per treating investigator's opinion, additional treatment is required for better correction or to maintain the results.

Clinical data were collected at all in clinic visits, including standardized facial photographs, pain perception self-assessement was recorded by subjects immediately after treatment. All subjects were asked for details of any Adverse Events (AEs) they had experienced. Subjects were asked to rate aesthetic results and Patient Satisfaction questionnaire at each follow-up visit. Physicians were asked to rate aesthetic results as well and details of the treatment session were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women, over the age of 18, seeking correction of facial wrinkles and folds and/or soft tissue augmentation.
* Subjects who are willing and able to read, understand and sign informed consent.

Exclusion Criteria:

* Subjects with known contraindications to the treatment (as per device IFU).
* Subjects considered to be unsuitable to participate, in the investigator's opinion, for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects over the age of 18 who are seeking correction of facial wrinkles and folds and/or soft tissue augmentation.
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2025-05-18 (Actual)

PRIMARY OUTCOMES:
1. The frequency of reported adveres events (number of participants who experienced each reported adverse event) 2. The severity of reported adverse events (1=mild, 2=moderate, 3=severe) | Up to 56 weeks after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Glyance Ltd, Lod, Israel

IPD SHARING:
Plan to Share IPD: No